CLINICAL TRIAL: NCT03479853
Title: Clinical, Meibographic and Interferometric Evaluation of Phlyctenular Keratitis in Children - MEIBO-ROSACEE
Acronym: MEIBO-ROSACEE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SDN_2017_26
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Ocular Rosacea; Keratoconjunctivitis; Meibomian Gland Dysfunction
Keywords: Ocular Rosacea; Keratoconjunctivitis; Meibomian Gland; Interferometry; Child
MeSH Terms: conditions — Rosacea; Keratoconjunctivitis; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases : suffering from ocular or oculo-cutaneous rosacea: Classic ophthalmologic examination with visual acuity measurement and slit lamp examination of both eyes and eyelids. Then, meibographic and interferometric evaluation of his two inferior eyelids with the Lipiview device.
  Interventions: Procedure: Ophthalmologic examination and meibographic and interferometric evaluation (Lipiview device)
- Witnesses: Without any present or past palpebral meibomian Gland Dysfunction
  Classic ophthalmologic examination with visual acuity measurement and slit lamp examination of both eyes and eyelids. Then, meibographic and interferometric evaluation of his two inferior eyelids with the Lipiview device.
  Interventions: Procedure: Ophthalmologic examination and meibographic and interferometric evaluation (Lipiview device)

INTERVENTIONS:
Procedure: Ophthalmologic examination and meibographic and interferometric evaluation (Lipiview device) — Classic ophthalmologic examination with visual acuity measurement and slit lamp examination of both eyes and eyelids. Then, meibographic and interferometric evaluation of his two inferior eyelids with the Lipiview device.

SUMMARY:
The aim of this study is to describe the clinical, meibographic and interferometric manifestations of phlyctenular keratitis in children.

DETAILED DESCRIPTION:
The investigators are conducting a monocentric, transversal, epidemiologic study. 100 patients should be included: 50 children suffering from ocular rosacea, and 50 children with no palpebral or Meibomian disease. Witnesses will be matched on the age of the cases.

Patient and controls will undergo a classic ophthalmologic examination with visual acuity measurement and slit lamp examination of both eyes and eyelids. Then, the child will go through a meibographic and interferometric evaluation of his two inferior eyelids. This evaluation is made by an optometrist with the Lipiview device, and lasts a few minutes.

ELIGIBILITY:
Inclusion Criteria:

* Recruited from a specialized ophthalmologic consultation Rothschild Ophthalmologic Foundation, Paris, France.
* Cases : suffering from ocular or oculo-cutaneous rosacea
* Witnesses : without any present or past palpebral or meibomian disease

Exclusion Criteria:

* Unable to achieve the meibographic and interferometric examination (Lipiview)

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 2 and 16 : Cases, suffering from ocular or oculo-cutaneous rosacea and Witnesses without any present or past palpebral or meibomian disease
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Clinical severity | Day of inclusion
  Clinical severity is determined with a composite score, by the presence of chalazia, corneal lesions, neovascularization, phlyctena, loss of vision, superficial keratitis, anterior and posterior keratitis, meibomitis, palpebral margin keratinization, lagophthalmos, long term use of azithromycin treatment, treatment by ciclosporin eyedrops, intense cutaneous or ocular symptoms, long time evolution of the disease.
Meibographic severity | Day of inclusion
  The meibographic severity is determined by the level of Meibomian gland atrophy, data obtained with the Lipiview
Interferometric severity | Day of inclusion
  The interferometric severity is evaluated by the thickness of the lipid layer tear film, data obtained with the Lipiview
Number of abortive blinks | Day of inclusion
  Number of abortive blinks during the Lipiview exam

CONTACTS AND LOCATIONS:
Overall Officials: Serge DOAN, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided